CLINICAL TRIAL: NCT00081926
Title: Gleevec Trial in Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571AUS177; US177; RIGHT Trial
Record Dates: First submitted 2004-04-26; First posted 2004-04-29 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; Chronic Myelogenous Leukemia; RIGHT Trial; US177; CSTI571
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Gleevec

SUMMARY:
This study will evaluate the molecular response to high dose Gleevec in newly diagnosed patients with Chronic Myelogenous Leukemia (CML) in Chronic Phase. This study will evaluate the ability of Gleevec to reduce the amount of abnormal protein that occurs in patients with CML.

Patients who are eligible to participate will be treated for 18 months. This trial will include male or female patients 18 years or older who are newly diagnosed (within 6 months) with CML.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Male or Female patients 18 years and older.
* Patient with a diagnosis of chronic myelogenous leukemia in chronic phase
* Within 6 months of initial diagnosis.
* Received any treatment for CML for less than 1 month prior to study entry with the exception of hydroxyurea and/or anagrelide.

Exclusion Criteria:

* Late chronic phase, accelerated phase or blastic phase
* Taking any other investigational agents within 28 days of starting the study
* If sibling donors have been identified and where allogeneic bone marrow transplantation will be the first line treatment.
* Another primary malignancy /cancer unless it is not considered clinically significant or does not require active intervention.
* If patients have heart problems or complications
* Pregnant or breast-feeding females
* Severe and/or uncontrolled disease such as diabetes, chronic renal disease, etc.
* Chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Diagnosis of human immunodeficiency virus (HIV) infection.
* Received any treatment for CML for longer than 1 month prior to study entry with the exception of hydroxyurea and/or anagrelide.
* Patient previously received radiotherapy to greater than 25% of the bone marrow.
* Patient had a major surgery within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2003-10; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis RIGHT Trial Hotline, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Cortes JE, Kantarjian HM, Goldberg SL, Powell BL, Giles FJ, Wetzler M, Akard L, Burke JM, Kerr R, Saleh M, Salvado A, McDougall K, Albitar M, Radich J; Rationale and Insight for Gleevec High-Dose Therapy (RIGHT) Trial Study Group. High-dose imatinib in newly diagnosed chronic-phase chronic myeloid leukemia: high rates of rapid cytogenetic and molecular responses. J Clin Oncol. 2009 Oct 1;27(28):4754-9. doi: 10.1200/JCO.2008.20.3869. Epub 2009 Aug 31. PMID 19720924
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com